CLINICAL TRIAL: NCT02423070
Title: Genome Transplant Dynamics
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915115; 15-H-N115
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Thoracic Organ Transplantation
Keywords: Cell-free DNA; Acute Rejection; Thoracic Organ Transplantation; Non-Invasive Testing; Chronic Rejection; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Heart and Lung Transplant patients

SUMMARY:
Study Description:

Heart and lung transplants can save lives, but long-term success is often limited by organ rejection that is hard to detect early. This study is testing a new, non-invasive blood test that looks for small pieces of DNA from the donor organ in the patient s blood. We believe higher levels of this donor DNA may signal early rejection before damage becomes permanent.

Hypothesis:

We believe that measuring donor-derived DNA in the blood can help detect early signs of rejection and improve outcomes for transplant patients.

The study also collects genetic and biological samples to explore why some people are more at risk of complications after transplant. This may help guide future research and treatments.

Who Can Join the Study:

People receiving a heart or lung transplant (or both), age 14 and older

People who are within three months of their transplant

People who can understand and agree to take part in the study

Participants will be asked to provide blood and other samples, and some of these will be used in lab research to explore new ideas about how and why transplant rejection happens.

This research could lead to better ways to monitor and treat patients after a heart or lung transplant - and help improve long-term survival and quality of life.

DETAILED DESCRIPTION:
Acute rejection (AR) occurs within the first 6 months after transplantation in 20 percent of heart- transplant patients and in 50 percent of lung-transplant patients. Given the often silent clinical presentation of AR, these patients require monitoring with repeated invasive and costly endomyocardial (EMB) or transbronchial biopsies (TBBx). Since organ transplantation is essentially genomic transplantation, our prior studies leveraged the use of distinctive graft and recipient genotype single-nuclear polymorphisms (SNPs) to barcode donor DNA circulating in recipient serum. We have shown that levels of donor DNA measured as the percentage of circulating donor-derived cell-free DNA (cfDNA) correlate with AR diagnosis and severity as detected by biopsy. The performance receiver operator curve (ROC) of cfDNA yielded an area under the curve (AUC) of 0.83. Using this technique, we can diagnose AR by measuring elevations in cfDNA up to 5 months before EMB-detected pathology. While these findings suggest that monitoring cfDNA may offer a high-performing, non-invasive, and early diagnostic tool of AR, further validation studies are required to determine its clinical utility. The ability to diagnose AR earlier than is possible with a biopsy offers an opportunity to investigate the pathogenesis of rejection as well as to identify potential AR biomarkers. Thus, the primary objective of this study is to validate the predictive accuracy and ROC characteristics of cfDNA for AR in a multicenter, prospective cohort study of heart and lung transplant patients, recruited through a consortium of 5 transplant centers in Washington, DC metropolitan area. The secondary objective is to determine the association between early graft injury caused by acute rejection and infection and the development of chronic rejection, i.e., chronic lung allograft dysfunction (CLAD) or chronic allograft vasculopathy (CAV). The exploratory objectives are: 1) to compare cfDNA characteristics in AMR (antibody-mediated rejection) and ACR (acute cellular rejection), 2) to study early immunological changes associated with a significant rise in cfDNA, and 3) to examine changes in microbiome architecture and other cell-free nucleic acids in rejection, 4) to determine if cfDNA trends correlate with treatment response for transplant complications, 5) to determine if the level of pre-transplant cfDNA identify patients at high risk of rejection post-transplant, 6) to determine genetic variants associated with post-transplant risk of rejection, high cfDNA levels and other complications.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Lung and heart transplant candidates. Dual organ transplants such as those that include lung or heart PLUS any other organ are also considered for enrollment.
* Subjects who have undergone lung or heart transplants and are within 3 months of transplantation.
* 14 years and older
* Able to understand and be willing to sign the informed consent form. Subjects undergoing a double transplant will sign a single consent.
* Retransplant candidates will be considered as a new transplants. These subjects will be approached for enrollment and if they consent to participate, they will be assigned a different SSPIN.

EXCLUSION CRITERIA:

-Pregnancy

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung and heart transplant candidates. Dual organ transplants such as those that include lung or heart PLUS any other organ are also considered for enrollment. -Subjects who have undergone lung or heart transplants and are within 3 months of transplantation. -14 years and older- Able to understand and be willing to sign the informed consent form. Subjects undergoing a double transplant will sign a single consent.- Retransplant candidates will be considered as a new transplants. These subjects will be approached for enrollment and if they consent to participate, they will be assigned a different SSPIN.
Sampling Method: Non-Probability Sample
Enrollment: 991 (Estimated)
Dates: Start 2015-06-25 (Actual); Primary Completion 2034-11-30 (Estimated); Study Completion 2034-11-30 (Estimated)

PRIMARY OUTCOMES:
To validate the predictive accuracy and ROC characteristics of circulating cell- free donor derived DNA (cfDNA) in multicenter, prospective cohort study of heart and lung transplant patients, recruited through a consortium of 5 transplant center... | At the time of biopsy-proven rejection
  Fold change in cfDNA at the time of biopsy-proven rejection

SECONDARY OUTCOMES:
To determine the association between early graft injury caused by acute rejection and infection and the development of chronic rejection, ie.,chronic lung allograft dysfunction (CLAD) or chronic allograft vasculopathy (CAV). | End of Study
  cfDNA in rejection grades 1R, 2R, and 3R, cfDNA at 1 month before biopsy diagnosis of AR, cfDNA after treatment of AR, cfDNA in ACR and AMR, spirometry grade of CLAD, angiographic grade of CAV, and number of AR per year, severity grade of clinically determined graft dysfunction, mean (cfDNA), all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Sean T Agbor-Enoh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (6):
- United States (6):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - INOVA Fairfax Medical, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known.

REFERENCES:
- [Background] Angelini A, Andersen CB, Bartoloni G, Black F, Bishop P, Doran H, Fedrigo M, Fries JW, Goddard M, Goebel H, Neil D, Leone O, Marzullo A, Ortmann M, Paraf F, Rotman S, Turhan N, Bruneval P, Frigo AC, Grigoletto F, Gasparetto A, Mencarelli R, Thiene G, Burke M. A web-based pilot study of inter-pathologist reproducibility using the ISHLT 2004 working formulation for biopsy diagnosis of cardiac allograft rejection: the European experience. J Heart Lung Transplant. 2011 Nov;30(11):1214-20. doi: 10.1016/j.healun.2011.05.011. Epub 2011 Aug 3. PMID 21816625
- [Background] De Vlaminck I, Khush KK, Strehl C, Kohli B, Luikart H, Neff NF, Okamoto J, Snyder TM, Cornfield DN, Nicolls MR, Weill D, Bernstein D, Valantine HA, Quake SR. Temporal response of the human virome to immunosuppression and antiviral therapy. Cell. 2013 Nov 21;155(5):1178-87. doi: 10.1016/j.cell.2013.10.034. PMID 24267896
- [Background] Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Deng MC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Elashoff B, Baron H, Yee J, Valantine HA; IMAGE Study Group. Gene-expression profiling for rejection surveillance after cardiac transplantation. N Engl J Med. 2010 May 20;362(20):1890-900. doi: 10.1056/NEJMoa0912965. Epub 2010 Apr 22. PMID 20413602
- [Derived] Goldberg JF, Bagchi P, Mercado A, Shah KB, Najjar SS, Tchoukina I, Rodrigo ME, Hsu S, Jang M, Kong H, Marboe CC, Berry GJ, Valantine HA, Agbor-Enoh S, Shah P; GRAfT Investigators. Identification of Heart Transplant Rejection Subtypes With Circulating MicroRNAs. Circ Heart Fail. 2026 Jan 12:e013141. doi: 10.1161/CIRCHEARTFAILURE.124.013141. Online ahead of print. PMID 41521923
- [Derived] Shah P, Agbor-Enoh S, Lee S, Andargie TE, Sinha SS, Kong H, Henry L, Park W, McNair E, Tchoukina I, Shah KB, Najjar SS, Hsu S, Rodrigo ME, Jang MK, Marboe C, Berry GJ, Valantine HA; GRAfT Investigators. Racial Differences in Donor-Derived Cell-Free DNA and Mitochondrial DNA After Heart Transplantation, on Behalf of the GRAfT Investigators. Circ Heart Fail. 2024 Apr;17(4):e011160. doi: 10.1161/CIRCHEARTFAILURE.123.011160. Epub 2024 Feb 20. PMID 38375637
- [Derived] Keller MB, Tian X, Jang MK, Meda R, Charya A, Berry GJ, Marboe CC, Kong H, Ponor IL, Aryal S, Orens JB, Shah PD, Nathan SD, Agbor-Enoh S. Higher Molecular Injury at Diagnosis of Acute Cellular Rejection Increases the Risk of Lung Allograft Failure: A Clinical Trial. Am J Respir Crit Care Med. 2024 May 15;209(10):1238-1245. doi: 10.1164/rccm.202305-0798OC. PMID 38190701
- [Derived] Keller M, Bush E, Diamond JM, Shah P, Matthew J, Brown AW, Sun J, Timofte I, Kong H, Tunc I, Luikart H, Iacono A, Nathan SD, Khush KK, Orens J, Jang M, Agbor-Enoh S. Use of donor-derived-cell-free DNA as a marker of early allograft injury in primary graft dysfunction (PGD) to predict the risk of chronic lung allograft dysfunction (CLAD). J Heart Lung Transplant. 2021 Jun;40(6):488-493. doi: 10.1016/j.healun.2021.02.008. Epub 2021 Feb 20. PMID 33814284
- [Derived] Agbor-Enoh S, Shah P, Tunc I, Hsu S, Russell S, Feller E, Shah K, Rodrigo ME, Najjar SS, Kong H, Pirooznia M, Fideli U, Bikineyeva A, Marishta A, Bhatti K, Yang Y, Mutebi C, Yu K, Kyoo Jang M, Marboe C, Berry GJ, Valantine HA; GRAfT Investigators. Cell-Free DNA to Detect Heart Allograft Acute Rejection. Circulation. 2021 Mar 23;143(12):1184-1197. doi: 10.1161/CIRCULATIONAHA.120.049098. Epub 2021 Jan 13. PMID 33435695
- [Derived] Agbor-Enoh S, Chan JL, Singh A, Tunc I, Gorham S, Zhu J, Pirooznia M, Corcoran PC, Thomas ML, Lewis BGT, Jang MK, Ayares DL, Horvath KA, Mohiuddin MM, Valantine H. Circulating cell-free DNA as a biomarker of tissue injury: Assessment in a cardiac xenotransplantation model. J Heart Lung Transplant. 2018 Aug;37(8):967-975. doi: 10.1016/j.healun.2018.04.009. Epub 2018 Apr 26. PMID 29933912
- [Derived] Agbor-Enoh S, Jackson AM, Tunc I, Berry GJ, Cochrane A, Grimm D, Davis A, Shah P, Brown AW, Wang Y, Timofte I, Shah P, Gorham S, Wylie J, Goodwin N, Jang MK, Marishta A, Bhatti K, Fideli U, Yang Y, Luikart H, Cao Z, Pirooznia M, Zhu J, Marboe C, Iacono A, Nathan SD, Orens J, Valantine HA, Khush K. Late manifestation of alloantibody-associated injury and clinical pulmonary antibody-mediated rejection: Evidence from cell-free DNA analysis. J Heart Lung Transplant. 2018 Jul;37(7):925-932. doi: 10.1016/j.healun.2018.01.1305. Epub 2018 Jan 31. PMID 29500138